CLINICAL TRIAL: NCT06807970
Title: Novel Perioperative Optimization of Obese Osteoarthritic Patients Pending Total Knee Replacement With Glucagon-like Peptide-1 Receptor Agonist (NPO-OOPS-TKR)
Brief Title: Optimization of Obesity for Total Knee Replacement With Glucagon-like Peptide-1 Receptor Agonist
Acronym: NPO-OOPS-TKR
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Lawrence Lau, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW24-423
Record Dates: First submitted 2025-01-15; First posted 2025-02-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GLP-1RA (Experimental): Intervention group: GLP-1RA +TKR:
  Patients in intervention group will have GLP-1RA semaglutide for 48 weeks and then stops for one month before and after TKR following the latest anesthesia guideline for GLP-1RA. Followed by TKR They will continue semaglutide for 48 weeks during the post-operative follow-up period. This is decided based on balancing treatment effect of semaglutide, waiting time for TKR, and TKR follow-up requirement. In Hong Kong, waiting time for TKR would be ~4 years and so a period of 12 months treatment of semaglutide is reasonable. And in the STEP 6 trial, weight loss at week 52 (-12%) is similar to that in study end at week 68(-13·2%), and STEP5 trial showed maintaining semaglutide to week 104 could maintain weight loss of similar degree as in week 52. And the consensus of assessing TKR Patient-Reported Outcome Measures (PROMs) is one year follow up.
  Interventions: Drug: Glucagon-like peptide-1 receptor agonists (GLP 1 RA)
- Control (standard treatment) (Placebo Comparator): Control Group: TKR alone:
  If patients are randomized to the control group, they will receive routine follow-up with general advice on diet and physical activity but will not receive semaglutide, and will not be offered a specific management program for their weight. This is in line with current practice.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Drug: Glucagon-like peptide-1 receptor agonists (GLP 1 RA) — Patients in intervention group will have GLP-1RA semaglutide for 48 weeks and then stops for one month before and after TKR following the latest anesthesia guideline for GLP-1RA. Followed by TKR They will continue semaglutide for 48 weeks during the post-operative follow-up period. This is decided based on balancing treatment effect of semaglutide, waiting time for TKR, and TKR follow-up requirement. In Hong Kong, waiting time for TKR would be ~4 years and so a period of 12 months treatment of semaglutide is reasonable. And in the STEP 6 trial, weight loss at week 52 (-12%) is similar to that in study end at week 68(-13·2%), and STEP5 trial showed maintaining semaglutide to week 104 could maintain weight loss of similar degree as in week 52. And the consensus of assessing TKR Patient-Reported Outcome Measures (PROMs) is one year follow up.
  Arms: GLP-1RA
Other: Control (Standard treatment) — If patients are randomized to the control group, they will receive routine follow-up with general advice on diet and physical activity but will not receive semaglutide, and will not be offered a specific management program for their weight. This is in line with current practice.
  Arms: Control (standard treatment)

SUMMARY:
Studies have shown that obese patients undergoing total knee replacement (TKR) surgery face a higher risk of perioperative issues such as increased use of pain medication, surgical site infections, and the need for revision surgeries compared to non-obese patients. Obesity is also linked to more significant preoperative pain and lingering symptoms post-surgery. Consequently, there's a growing interest in weight loss interventions prior to TKR to enhance perioperative care and outcomes. Recent retrospective studies have indicated that such interventions can improve physical function post-TKR.

Research focusing on weight loss interventions before joint replacement surgery is limited.

There is currently a gap in research regarding RCTs on weight loss interventions using anti-obesity drugs before TKR, particularly in Asian populations.

One promising avenue under exploration involves the use of glucagon-like peptide 1 receptor agonists (GLP-1RAs) as anti-obesity medication before total knee replacement (TKR) surgery. However, there are currently no randomized controlled trials (RCTs) examining the effects of GLP-1RAs on knee arthroplasty outcomes. Large database studies have indicated that GLP-1RAs may decrease the likelihood of certain post-surgery complications but increase the risk of others.

In summary, addressing obesity through weight loss interventions, particularly with GLP-1RAs, holds promise for improving outcomes in TKR patients. However, further research, including randomized controlled trials, is necessary to fully understand the effects of GLP-1RAs on perioperative outcomes and patient health.

DETAILED DESCRIPTION:
2.1 Hypothesis Hypothesis for this pilot trial is conducting trial of GLP-1RA for perioperative optimization for TKR feasible. The null hypothesis for the full trial is that clinical, functional and quality of life (QoL) outcomes in obese patients undergoing TKR will not be improved if this is preceded by GLP-1 RA induced weight loss.

3. Study objective The primary aims of this pilot study are 1) estimate adherence, tolerability and follow-up rates, 2) recruitment and management challenges.

The secondary aims are to assess the effect of semaglutide for perioperative optimization in TKR and gather data to estimate the feasibility like tolerability and sample size for a future trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years old
* BMI ≥27 kg/m2
* On the surgical waiting list for primary TKR
* Willing and able to cooperate in a weight management programme.
* Meeting indication for semaglutide

Exclusion Criteria:

* Revision surgery or surgery for neoplastic disease
* A medical condition which in the opinion of the investigators makes the patient unsuitable for participation in the trial
* Contraindication to GLP-1RA, like history of pancreatitis, severe gastrointestinal diseases such as gastroparesis, thyroid cancer, and inflammatory bowel disease
* Lack of acceptance of the randomisation process.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  Assess at enrolment, prior to and after TKR, and at each follow-up till 12 months. Pain is chosen as the primary outcome because up to 14 patients in weight loss groups (versus 2 patients in control groups) in previous studies chosen to decline/delay TKR due to pain relief, suggesting a prominent effect of weight optimization on pain relief.
  Pain is evaluated using two approaches. The first method is visual analog scale which involves the numeric rating scale, which ranges from 0 to 10, with 0 representing no pain and 10 representing the most intense pain. The second method involves monitoring analgesic consumption, with higher consumption indicating more severe pain.

SECONDARY OUTCOMES:
A composite score of clinical situation | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  A patient is likely to have a composite score reported in numerical scale if they experience the following conditions:
  (i) Failed same-day rehabilitation (within 24 hours) (ii) Have any peri-operative complications (medical or surgical) (iii) Have any post-operative complications (medical or surgical) leading to delayed discharge, such as fractures, neuropraxia, sepsis, nosocomial infections, myocardial infarction, bowel obstruction, venous thromboembolism, cardiovascular events, or renal failure (iv) Have any wound complications (breakdown, infections, hematomas, dehiscence) (v) Have joint infections as per Musculoskeletal Infection Society (MSIS) Criteria (vi) Have any unplanned procedures and/or readmissions within the first 12 months following total knee replacement (TKR) (vii) Death from any cause
  A higher composite score suggests that the patients are in a poorer condition.
Length of stay | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  Patients' conditions worsen as the length of stay (unit in day) in acute and rehabilitation hospitals for total knee replacement (TKR), as well as any subsequent related admissions, increases.
Body weight | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  Body weight (kg - kilogram) will be measured at each visit.
Radiological parameters | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  Lower limb alignment will be measured in degree to assess changes before and after surgery.
height | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  height (cm-centimètre)will be measured at each visit.
waist circumference | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  waist circumference (cm - centimètre) will be measured at each visit.
blood pressure | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  Both systolic and diastolic blood pressure (mmHg - Millimeter of mercury) will be measured at each visit.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) consists of 24 items divided into 3 subscales Pain (5 items), Stiffness (2 items)Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total WOMAC score.
The Knee Society Score | As part of the standard of care when undergoing TKR, patients are routinely assessed at enrolment, 1 month and same day before surgery, and at 6 weeks,3 months, 6 months and 12 months post-surgery.
  The Knee Society Score is clinician-administered consisting of a Knee and Function Score. The Knee Score rates the knee joint itself and allocates a maximum of 100 points for the evaluation of range of motion (1 point per 5°, maximum 125°), stability (medial/lateral (15 points) and anterior/posterior (10 points)) and pain (50 points) with deductions for extension lag, flexion contracture and malalignment (if leg axis < 5 or > 10° on radiological examination) [1]. A maximum score of 100 points represents a well-aligned knee with 125° of motion, almost none anteroposterior or mediolateral instability and no pain. The Function Score considers walking distance (50 points) and stair climbing (50 points) with deduction for the use of a walking aid . A patient who can walk unlimited and has no trouble with climbing stairs will obtain the maximum Function Score of 100 points.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lau, FRCS, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
for further patient privacy protection